CLINICAL TRIAL: NCT01595503
Title: Functional Targeting of Transcranial Magnetic Stimulation for the Treatment of Refractory Auditory Hallucinations in Schizophrenia
Brief Title: Transcranial Magnetic Stimulation for the Treatment of Auditory Hallucinations in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00046254
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, auditory hallucination
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fMRI-based targeting (Experimental)
  Interventions: Procedure: rTMS with fMRI-based targeting
- landmark-based targeting (Active Comparator)
  Interventions: Procedure: rTMS with landmark-based targeting

INTERVENTIONS:
Procedure: rTMS with fMRI-based targeting — Inhibitory (low frequency) 1-Hz rTMS will be applied to the secondary auditory cortex during 10 daily 20-minute treatment sessions. An fMRI scan combined with a language task will be used to localize the secondary auditory cortex, followed by neuronavigation to identify the scalp location overlying the targeted cortex.
  Arms: fMRI-based targeting
Procedure: rTMS with landmark-based targeting — Inhibitory (low frequency) 1-Hz rTMS will be applied over the left temporoparietal cortex (TPC) during 10 daily 20-minute treatment sessions, with the stimulating coil located midway between the left temporal (T3) and parietal (P3) scalp landmarks, using the International 10-20 system for EEG.
  Arms: landmark-based targeting

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a new noninvasive therapy that uses magnetic energy applied to the scalp to modulate activity in the underlying regions of the brain. In this study we will examine the efficacy of treating auditory hallucinations in schizophrenia with rTMS, comparing two methods to target stimulation to a language processing region of the brain. One method targets the stimulation site using scalp landmarks, while the other uses functional magnetic resonance imaging (fMRI) combined with a language task.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Male or female, aged 18 to 60
* Willing to comply with all study procedures and be available for the duration of the study
* Primary diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV (29)
* Currently reporting AHs, rated a minimum of 4 (moderate) on the auditory hallucination item of the Brief Psychiatric Rating Scale (BPRS; 27), and AH will be present daily
* AHs must have failed to resolve after a minimum of two adequate trials (doses within standard therapeutic range for a minimum of 8 weeks each) of psychotropic medication including at least one atypical antipsychotic medication; documented trials of antipsychotic medication limited by intolerable side effects, e. g. extra-pyramidal symptoms, tardive dyskinesia, weight gain, neuroleptic-induced dysphoria, will also be considered as equivalent to adequate trials.
* Weight and girth compatible with the bore of the MRI scanner; generally men over 6 feet tall < 250 lbs, men under 6 feet tall < 220 lbs, women over 5'11" tall < 220 lbs, or women under 5'10" tall < 200 lbs

Exclusion Criteria:

* Substance abuse or dependence in the past 1 month
* Current or past history of serious medical or neurological illness that could compromise brain function or present an increased risk of seizure, e. g. conditions that may significantly alter electrolyte balance, stroke, epilepsy, any history of seizure;
* Pregnant or trying to become pregnant;
* Inability to tolerate small, enclosed spaces without anxiety;
* Metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition, e. g. aneurysm clips, retained particles, neurostimulators, foil-backed transdermal patches;
* Facial tattoos with metallic ink
* Inability to follow study protocol
* Change in antipsychotic therapy in previous 2 weeks
* Currently under an alternative treatment order
* Unstable symptoms which could, in the judgment of the study team, exhibit symptomatic worsening over the course of the protocol
* Current treatment with another investigational drug or other intervention
* Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study;
* No quantifiable motor threshold such that TMS dosage cannot be accurately determined

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan F Taylor, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Psychiatry Depression Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated because of the small enrollment (2 or 3 subjects per treatment arm), the data that was examined was pooled for all the subjects. At the time of results reporting it is impossible to disambiguate the two arms. Randomization tables are not available; hence, we cannot report the results by treatment arm.
Groups:
- rTMS With Either fMRI-based Targeting or Landmark Based Targeting.: rTMS Inhibitory (low frequency) 1-Hz rTMS will be applied to the secondary auditory cortex during 10 daily 20-minute treatment sessions.
Period: Overall Study
Arm/Group | rTMS With Either fMRI-based Targeting or Landmark Based Targeting.
Started | 5
Completed (Study was discontinued because of poor recruitment and insufficient data for analysis) | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- rTMS With fMRI-based Targeting or Landmark Based Targeting: rTMS: Inhibitory (low frequency) 1-Hz rTMS will be applied to the secondary auditory cortex during 10 daily 20-minute treatment sessions.
Arm/Group | rTMS With fMRI-based Targeting or Landmark Based Targeting
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Auditory Hallucinations
Description: Hallucination Change Scale (Hoffman RE, Gueorguieva R, Hawkins KA, Varanko M, Boutros NN, Wu YT, et al. (2005): Temporoparietal transcranial magnetic stimulation for auditory hallucinations: safety, efficacy and moderators in a fifty patient sample. Biol Psychiatry. 58:97-104.) Baseline score, by definition: 10 Range: 0 (no hallucinations) to 20 (hallucinations twice as bad as baseline) Thus, a score of less than 10 means that hallucinations were reduced, whereas a score of greater than 10 means that hallucinations were increased.
Time Frame: Two weeks
Population: The two original groups: with fMRI targeted and landmark based were planned to be analyzed separately, the data available at the time of results reporting, is no longer separable. Thus all treated participants are included in a single arm. While this does not allow comparison between the two approaches to rTMS usage, it still allows one to see the impact of using rTMS with one method or the other, albeit still in a tiny sample size.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- rTMS: rTMS : Inhibitory (low frequency) 1-Hz rTMS will be applied to the secondary auditory cortex during 10 daily 20-minute treatment sessions.
Arm/Group | rTMS
Number analyzed (Participants) | 5
score on a scale | 5.9 (1.7)

ADVERSE EVENTS:
Arm/Group | rTMS
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes